CLINICAL TRIAL: NCT00072514
Title: A Phase II Study Evaluating the Efficacy of Gemcitabine, Carboplatin, and Dexamethasone and Rituximab for Previously Treated Lymphoid Malignancies
Brief Title: Gemcitabine Hydrochloride, Carboplatin, Dexamethasone, and Rituximab in Treating Patients With Previously Treated Lymphoid Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ajay Gopal, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSOC 2003; NCI-2011-00035 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2003-11-04; First posted 2003-11-05 (Estimated); Results first posted 2017-06-29 (Actual); Last update posted 2017-06-29 (Actual); Status verified 2017-05

CONDITIONS: Adult Nasal Type Extranodal NK/T-cell Lymphoma; Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Cutaneous B-cell Non-Hodgkin Lymphoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Hepatosplenic T-cell Lymphoma; Intraocular Lymphoma; Nodal Marginal Zone B-cell Lymphoma; Noncutaneous Extranodal Lymphoma; Peripheral T-cell Lymphoma; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Small Lymphocytic Lymphoma; Small Intestine Lymphoma; Splenic Marginal Zone Lymphoma; Testicular Lymphoma; Waldenstrom Macroglobulinemia
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Intraocular Lymphoma; Lymphoma, B-Cell, Marginal Zone; Lymphoma, T-Cell, Peripheral; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia | interventions — Gemcitabine; Carboplatin; Dexamethasone; Calcium Dobesilate; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Patients receive gemcitabine hydrochloride intravenously (IV) over 30 minutes on days 1 and 8, carboplatin IV over 30-60 minutes on day 1, and dexamethasone orally (PO) on days 1-4. Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity. Patients with CD20-POSITIVE LYMPHOMAS also receive rituximab IV on day 8.
  Interventions: Drug: gemcitabine hydrochloride; Drug: carboplatin; Drug: dexamethasone; Biological: rituximab

INTERVENTIONS:
Drug: gemcitabine hydrochloride — Given IV
  Other Names: dFdC; difluorodeoxycytidine hydrochloride; gemcitabine; Gemzar
Drug: carboplatin — Given IV
  Other Names: Carboplat; CBDCA; JM-8; Paraplat; Paraplatin
Drug: dexamethasone — Given PO
  Other Names: Aeroseb-Dex; Decaderm; Decadron; DM; DXM
Biological: rituximab — Given IV in CD20-POSITIVE LYMPHOMAS cases
  Other Names: IDEC-C2B8; IDEC-C2B8 monoclonal antibody; Mabthera; MOAB IDEC-C2B8; Rituxan

SUMMARY:
This pilot phase II trial studies the side effects and how well giving gemcitabine hydrochloride, carboplatin, dexamethasone, and rituximab together works in treating patients with previously treated lymphoid malignancies. Drugs used in chemotherapy, such as gemcitabine hydrochloride, carboplatin, and dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Giving more than one drug (combination chemotherapy) and giving monoclonal antibody therapy with chemotherapy may kill more cancer cells

DETAILED DESCRIPTION:
OBJECTIVES:

I. To determine the feasibility and safety of Gemcitabine/Carboplatin/Dexamethasone with or without Rituximab in previously treated lymphoid malignancies (rituximab will only be evaluated in CD20 positive malignancies).

II. To determine the efficacy of the above regimen.

III. To determine the ability to proceed to blood stem peripheral blood collection following the above regimens (the impact of above regimen on stem cell reserve).

IV. To determine remission duration.

All patients are treated with gemcitbine, carboplatin, and dexamethasone. Patients with CD20 + lymphomas also receive rituximab.

After completion of study treatment, patients are followed up at 3-4 weeks and then every 6 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have relapsed or primary refractory lymphoid malignancy (including B-cell, T-cell, or Hodgkin's Disease)
* Revised European American classification (REAL), or World Health Organization (WHO) classification of patients malignancies must be provided
* Patients must have measurable disease defined as lesions that can be accurately measured in two dimensions by computed tomography (CT), magnetic resonance imaging (MRI), medical photograph (skin or oral lesion), plain x-ray, or other conventional technique and a greatest transverse diameter of 1 cm or greater; or palpable lesions with both diameters >= 2 cm; Note: CT scans remain the standard for evaluation of nodal disease
* Patients must have a bone marrow aspirate and biopsy within 28 days of enrollment and no intervening anticancer therapy
* Patients must have a CT of chest, abdomen, and pelvis within 28 days of enrollment; patients with evidence of adenopathy in the neck must have a CT of neck
* Patients should not have evidence active central nervous system lymphoma
* Patients must have a Southwest Oncology Group (SWOG) performance status of 0, 1, or 2
* Patients should have absolute neutrophil count (ANC) >= 1,500/uL; exception: patients with cytopenia thought to be due to disease in their bone marrow, that do not meet this criteria, may be enrolled on the protocol at the Study Chair's discretion
* Patients should have platelets >= 100,000/uL; exception: patients with cytopenia thought to be due to disease in their bone marrow, that do not meet this criteria, may be enrolled on the protocol at the Study Chair's discretion
* Serum bilirubin less than 2 times the upper limit of normal
* Serum creatinine less than 1.5 times the upper limit of normal and creatinine clearance greater than 50/ mL per minute
* Patients must have serum lactate dehydrogenase (LDH) performed within 14 days prior to treatment
* All patients must be informed of the investigational nature of this study and have given written consent in accordance with institutional and federal guidelines
* Must anticipate that patient will complete at least 2 cycles of chemotherapy

Exclusion Criteria:

* Patients known to be human immunodeficiency virus (HIV) positive
* Pregnant or nursing women; men or women of reproductive potential may not participate unless they have agreed to use an effective contraceptive method
* Patients with other prior malignancies except for adequately treated basal cell carcinoma, squamous cell carcinoma of the skin, cervical cancer in situ, or other cancer from which the patient has been disease-free for 5 years or greater unless approved by the Principal Investigator (PI)
* Patients that are refractory (i.e., not responded or progressed within 6 months) to a carboplatin or cisplatin-based regimen or a gemcitabine-based regimen
* Patients with active hepatitis B virus (HBV) infection or hepatitis
* Patients that have other medical conditions that would contraindicate treatment with aggressive chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2003-08; Primary Completion 2008-07 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Gopal, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment
Started | 55
Completed | 51
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 51
Age, Continuous [Median (Full Range); unit: years] | 58 [19 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 30

OUTCOME MEASURES:

1. Primary Outcome: Ability to Successfully Deliver the Investigational Therapy Without Incurring the Protocol Suspension Rules
Description: Count of participants that received the investigational therapy without incurring the protocol suspension rules. A stopping rule for safety was employed such that the study would be suspended if sufficient evidence indicated that the true grade 4-5 non-hematologic toxicity rate exceeded 10%.
Time Frame: At 3-4 weeks after completion of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 51
Participants | 51

2. Secondary Outcome: Overall and Complete Response Rates
Description: Response was assessed per standard criteria (Cheson BD, Horning SJ, Coiffier B, et al. Report of an international workshop to standardize response criteria fornon-Hodgkin's lymphomas. J Clin Oncol 1999;17:1244-1253.)
Time Frame: 3-4 weeks after completion of study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment
Number analyzed (Participants) | 51
percentage of participants
  Overall | 67 [54 to 80]
  Complete | 31 [19 to 44]

3. Secondary Outcome: Hematologic and Non-hematologic Adverse Events.
Description: Count of participants with grade 3/4 hematologic and non-hematologic adverse events.
Time Frame: 3-4 weeks after completion of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 51
Participants
  Hematologic Grade 3 | 10
  Hematologic Grade 4 | 39
  Non-Hematologic Grade 3 | 23
  Non-Hematologic Grade 4 | 2

4. Secondary Outcome: Peripheral Blood Stem Cell Collection
Description: Count of patients that attempted and had successful autologous peripheral blood stem cell (PBSC) collection.
Time Frame: Up to 12 weeks
Population: Successful PBSC collection is only considered in those patients that attempted PBSC collection.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 51
Participants
  Attempted PBSC Collection | 17
  Successful PBSC Collection: number analyzed (Participants) | 17
  Successful PBSC Collection | 17

ADVERSE EVENTS:
Arm/Group | Treatment
Serious Adverse Events (participants affected / at risk) | 0/51
Other Adverse Events (participants affected / at risk) | 45/51
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=51)
Neutrophils (Blood and lymphatic system disorders) | 38
Hemoglobin (Blood and lymphatic system disorders) | 18
Hemorrhage (Blood and lymphatic system disorders) | 5
Infection (Infections and infestations) | 12
Platelets (Blood and lymphatic system disorders) | 45
Thromboses (Blood and lymphatic system disorders) | 3
Hypotension (Vascular disorders) | 3
Constitutional (General disorders) | 5
GI (Gastrointestinal disorders) | 4
Matabolic/Laboratory (Metabolism and nutrition disorders) | 11
Neurology (Nervous system disorders) | 3
Pain (General disorders) | 6
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes